CLINICAL TRIAL: NCT06988800
Title: A Randomized Controlled Trial Examining the Impact of a Guided Paced Breathing Audiovisual Intervention on Psychosocial Functioning in Palestinian Adolescents
Brief Title: Musically-Guided Paced Breathing Improves Mental Health in War-Affected Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muvik Labs (Industry)
Collaborators: MECI (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MECI_Adolescent
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Anxiety; Self-Efficacy; Depression Not Otherwise Specified
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Guided Paced Breathing Audiovisual Intervention (Experimental): Paced Breathing intervention delivered
  Interventions: Device: Paced breathing wellness breathing sessions
- Guided Mindfulness Audiovisual Intervention (Experimental): Mindfulness intervention delivered
  Interventions: Device: Mindfulness video sessions
- Control (No Intervention): Participants in the control condition completed other typical after-school activities while participants in the intervention condition completed one of two breathing interventions: paced breathing (paced), or mindful breathing (mindfulness). Participants in the control condition were given the opportunity to complete the intervention after the study ended.

INTERVENTIONS:
Device: Paced breathing wellness breathing sessions — The paced breathing condition used timed auditory and visual cues to guide participants through breathing cycles at a rate of five breaths per minute, designed to stimulate the parasympathetic nervous system and promote relaxation. The audiovisual cues included spoken instructions, music, and breath-like sounds. The tonal audio cues rose in pitch during inhalation and fell during exhalation, creating a clear auditory signal for breath pacing. The same harmonic drone used in the mindfulness intervention provided a calming background, though here it was combined with the rhythmic pacing. Visually, the pacing was synchronized with the image of a lotus flower opening during inhalation and closing during exhalation, reinforcing the breathing rhythm.
  Arms: Guided Paced Breathing Audiovisual Intervention
Device: Mindfulness video sessions — The audio component of the mindfulness intervention featured a female narrator guiding participants through mindfulness exercises, focusing on breath awareness and cultivating non-judgmental attention to thoughts and feelings. Ambient tonal sounds, including a harmonic drone with slow timbral changes, played softly in the background to support relaxation. Importantly, no rhythmic audio cues were included to avoid inducing breathing entrainment. This setup emphasized passive, mindful observation rather than active breath control, encouraging participants to observe their bodily sensations and thoughts without judgment.
  Arms: Guided Mindfulness Audiovisual Intervention

SUMMARY:
Examine the impact of a mindfulness condition, a guided paced breathing audiovisual intervention condition, and a guided paced breathing audiovisual intervention plus take-home application condition compared to a matched control condition on anxiety symptoms.

DETAILED DESCRIPTION:
Methodology:

Sample and population

Individuals will be eligible if they attend the after-school program in Palestine through the Middle East Children's Institute (MECI) and are in grades 9-12. The MECI after school program is a free enrichment service provided to Palestinian youth at no charge. The activities include healthy meals, psychosocial support, creative art, sports, and drama.

Study setting The Middle East Children's Institute after-school program in Palestine.

Recruitment All eligible adolescents will be given information about the study (including that it is optional and voluntary) and provided with a consent form to bring home to their parents. Study staff will follow-up with the families of potentially eligible adolescents up to three times to ask if they have questions about the study and/or to remind them to return the signed consent form if they would like to participate.

Study duration Each intervention will have 14 sessions, delivered 2 times a week for 5 weeks in a group format in school classrooms, and an additional 2 weeks following a one month Ramadan period with no intervention delivered. Each group will consist of approximately 10 adolescents, and each intervention will have a duration of approximately less than 10 minutes long. Multiple sessions will be necessary to complete all assessments before and after the intervention.

Data collection and tools

There will be several non-invasive survey instruments utilized in this study.

Demographics. At baseline, participants will complete an investigator-developed self-report questionnaire that asks about participant age and gender identity.

Anxiety. As the primary outcomes measure, participants will complete the Revised Children's Manifest Anxiety Scale (RCMAS) self-report questionnaire. The RCMAS lists 37 feelings or actions and participants respond "yes" if that item is typical of their own feelings/actions, or "no" if not. The RCMAS produces a total anxiety score and three subscales: physiological anxiety, worry/oversensitivity, and social concerns/concentration. The Arabic version of the RCMAS has shown to have acceptable reliability and validity in youth.

Self-Efficacy. As a secondary outcome measure, a translated version of the Self-Efficacy Questionnaire for Children (SEQ-C) will be used. The SEQ-C includes three 8-item scales that measure academic, social, and emotional self-efficacy. The academic self-efficacy scale includes questions about the person's perception of achieving academic goals. The social self-efficacy scale addresses social challenges, and the emotional self-efficacy scale includes questions about coping with unpleasant problems or events.

Depression. As a secondary outcome measure, depression will be measured by the translated PHQ (Patient Health Questionnaire) -9.

Incentives for participants

Participants will receive no financial or other compensation.

ELIGIBILITY:
Inclusion Criteria:

Participating in MECI after school program and between the ages of 13 and 17.

Exclusion Criteria:

Not participating in MECI after school program or outside of the ages of 13 and 17.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 213 (Actual)
Dates: Start 2024-01-21 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chelsea Gordon, PhD, Study Director — Muvik Labs
Locations (1):
- MECI, Deir Ghassaneh, West Bank, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] AlHadi AN, AlAteeq DA, Al-Sharif E, Bawazeer HM, Alanazi H, AlShomrani AT, Shuqdar RM, AlOwaybil R. An arabic translation, reliability, and validation of Patient Health Questionnaire in a Saudi sample. Ann Gen Psychiatry. 2017 Sep 6;16:32. doi: 10.1186/s12991-017-0155-1. eCollection 2017. PMID 28878812

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Students were included in this study if they were children aged 13-17 years and enrolled in January 2024 at a school in a war-torn area in the West Bank in the Middle East.
Period: Intervention Period 1 - 5 Weeks
Arm/Group | Guided Paced Breathing Audiovisual Intervention | Guided Mindfulness Audiovisual Intervention | Control
Started | 64 | 77 | 72
Completed | 64 | 77 | 72
Not Completed | 0 | 0 | 0
Period: Intervention Period 2 - 2 Weeks
Arm/Group | Guided Paced Breathing Audiovisual Intervention | Guided Mindfulness Audiovisual Intervention | Control
Started | 64 | 77 | 72
Completed | 64 | 77 | 72
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guided Paced Breathing Audiovisual Intervention | Guided Mindfulness Audiovisual Intervention | Control | Total
Number analyzed (Participants) | 64 | 77 | 72 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.81 (.99) | 13 (1.1) | 14.45 (.97) | 13.75 (1.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 38 | 112
  Male | 28 | 39 | 34 | 101
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Palestine | 64 | 77 | 72 | 213
Self-Efficacy Questionnaire for Children [Mean (Standard Deviation); unit: units on a scale] — As a secondary outcome measure, a translated version of the Self-Efficacy Questionnaire for Children (SEQ-C) will be used. The SEQ-C includes three 8-item scales that measure academic, social, and emotional self-efficacy. The academic self-efficacy scale includes questions about the person's perception of achieving academic goals. The social self-efficacy scale addresses social challenges, and the emotional self-efficacy scale includes questions about coping with unpleasant problems or events.
  The subscale totals are added for a total score, ranging from 0-72, with a higher score being a posi
  units on a scale | 56.67 (15.92) | 53.76 (19.4) | 54.9 (17.29) | 55.05 (17.64)
Patient Health Questionnaire-9 [Mean (Standard Deviation); unit: units on a scale] — A validated measure of depressive symptoms, consisting of nine items assessing the frequency of depressive symptoms over the past two weeks. The Patient Health Questionnaire-9 (PHQ-9) has demonstrated strong psychometric properties, including reliability and validity in clinical and non-clinical populations, including the translated Arabic version.
  Scores range from 0-27, with a higher score indicating more depressive symptoms.
  units on a scale | 10.62 (5.64) | 9.44 (6.57) | 10.09 (6.59) | 10.03 (6.29)
Revised Children's Manifest Anxiety Scale [Mean (Standard Deviation); unit: units on a scale] — As the primary outcomes measure, participants will complete the Revised Children's Manifest Anxiety Scale (RCMAS) self-report questionnaire. The RCMAS lists 37 feelings or actions and participants respond "yes" if that item is typical of their own feelings/actions, or "no" if not. The RCMAS produces a total anxiety score and three subscales: physiological anxiety, worry/oversensitivity, and social concerns/concentration. The Arabic version of the RCMAS has shown to have acceptable reliability and validity in youth.
  The score ranges from 0-37, with a higher score indicating greater anxiety.
  units on a scale | 17.61 (8.13) | 18.67 (8.73) | 17.64 (8.39) | 18 (8.41)

OUTCOME MEASURES:

1. Primary Outcome: Revised Children's Manifest Anxiety Scale (RCMAS)
Description: As the primary outcomes measure, participants will complete the Revised Children's Manifest Anxiety Scale (RCMAS) self-report questionnaire. The RCMAS lists 37 feelings or actions and participants respond "yes" if that item is typical of their own feelings/actions, or "no" if not. The RCMAS produces a total anxiety score and three subscales: physiological anxiety, worry/oversensitivity, and social concerns/concentration. The Arabic version of the RCMAS has shown to have acceptable reliability and validity in youth.
  The score ranges from 0-37, with a higher score indicating greater anxiety.
Time Frame: From enrollment to the end of treatment at 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guided Paced Breathing Audiovisual Intervention | Guided Mindfulness Audiovisual Intervention | Control
Number analyzed (Participants) | 64 | 77 | 72
units on a scale | 24.88 (6.61) | 26.2 (5.82) | 17.91 (8.28)
Statistical Analysis 1: Comparison: Guided Paced Breathing Audiovisual Intervention vs Guided Mindfulness Audiovisual Intervention vs Control; ANCOVAs and post hoc Tukey pairwise tests; Test type: Superiority; p < .001, ANCOVA; Odds Ratio (OR) = 37.1

2. Primary Outcome: Self-Efficacy Questionnaire for Children (SEQ-C)
Description: As a secondary outcome measure, a translated version of the Self-Efficacy Questionnaire for Children (SEQ-C) will be used. The SEQ-C includes three 8-item scales that measure academic, social, and emotional self-efficacy. The academic self-efficacy scale includes questions about the person's perception of achieving academic goals. The social self-efficacy scale addresses social challenges, and the emotional self-efficacy scale includes questions about coping with unpleasant problems or events.
  The subscale totals are added for a total score, ranging from 0-72, with a higher score being a positive indicator of greater self-efficacy.
Time Frame: From enrollment to the end of treatment at 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guided Paced Breathing Audiovisual Intervention | Guided Mindfulness Audiovisual Intervention | Control
Number analyzed (Participants) | 64 | 77 | 72
units on a scale | 64.81 (16.15) | 64.65 (14.97) | 49.7 (20.29)
Statistical Analysis 1: Comparison: Guided Paced Breathing Audiovisual Intervention vs Guided Mindfulness Audiovisual Intervention vs Control; ANCOVAs and post hoc Tukey pairwise tests; Test type: Superiority; p < .001, ANCOVA; Odds Ratio (OR) = 19.5

3. Primary Outcome: Patient Health Questionnaire 9 (PHQ-9)
Description: A validated measure of depressive symptoms, consisting of nine items assessing the frequency of depressive symptoms over the past two weeks. The PHQ-9 has demonstrated strong psychometric properties, including reliability and validity in clinical and non-clinical populations, including the translated Arabic version.
  Scores range from 0-27, with a higher score indicating more depressive symptoms.
Time Frame: From enrollment to the end of treatment at 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guided Paced Breathing Audiovisual Intervention | Guided Mindfulness Audiovisual Intervention | Control
Number analyzed (Participants) | 64 | 77 | 72
units on a scale | 5.82 (5.04) | 5.86 (5.71) | 10.83 (6.93)
Statistical Analysis 1: Comparison: Guided Paced Breathing Audiovisual Intervention vs Guided Mindfulness Audiovisual Intervention vs Control; ANCOVAs and post hoc Tukey pairwise tests; Test type: Superiority; p < .001, ANCOVA; Odds Ratio (OR) = 18.7

ADVERSE EVENTS:
Time Frame: From enrollment until one month after the final assessment was completed, up to 15 weeks.
Description: Adverse events (AEs) will be collected from the time of informed consent through the end of study participation. All AEs, regardless of severity or relationship to study intervention, will be documented with onset date, end date, severity (mild, moderate, severe), seriousness, causality (related or not related to study intervention), action taken, and outcome. AEs include software malfunction, participant pain or discomfort, physical or emotional, or any other health-related occurrence.
Arm/Group | Guided Paced Breathing Audiovisual Intervention | Guided Mindfulness Audiovisual Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/77 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/77 | 0/72
Other Adverse Events (participants affected / at risk) | 0/64 | 0/77 | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT06988800/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT06988800/ICF_001.pdf